CLINICAL TRIAL: NCT02648841
Title: A Randomized Phase III Study of Adjuvant Chemotherapy With or Without Chemo-radiotherapy in Patients With Local Advanced Gastric Cancer After D2 Resection.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Jin, M.D., M.D., Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2015 YL-02
Record Dates: First submitted 2016-01-04; First posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; adjuvant chemo-radiotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adjuvant Chemotherapy (Active Comparator): The interventions of adjuvant chemotherapy group is 8 cycles of SOX(S-1+Oxaliplatin) chemotherapy to be given. The SOX chemotherapy regimen is as follow: S-1 40-60mg Bid, Oral, D1-14, Q21D; Oxaliplatin 130mg/m2, ivgtt, D1, Q21d.
  Interventions: Drug: Adjuvant chemotherapy for active comparator group
- Adjuvant Chemo-radiotherapy (Experimental): The interventions of adjuvant chemo-radiotherapy group is concurrent chemo-radiotherapy to be give after 4-6 cycles of chemotherapy. Total dose of 45Gy is delivered by IMRT Radiotherapy technique. The concurrent chemotherapy regimen is as follow: S-1 40-60mg Bid, Oral. Six cycles of SOX chemotherapy to be given. The SOX chemotherapy regimen is as follow: S-1 40-60mg Bid, Oral, D1-14, Q21D; Oxaliplatin 130mg/m2, ivgtt, D1, Q21d.
  Interventions: Radiation: Adjuvant Concurrent Chemo-radiotherapy; Drug: Adjuvant chemotherapy for experimental group

INTERVENTIONS:
Radiation: Adjuvant Concurrent Chemo-radiotherapy — Adjuvant concurrent chemo-radiotherapy will be given to the patients in the Experimental group after 4-6 cycles of SOX chemotherapy. Total dose of 45Gy is delivered by IMRT Radiotherapy technique. The concurrent chemotherapy regimen is as follow: S-1 40-60mg Bid, Oral.
  Arms: Adjuvant Chemo-radiotherapy
Drug: Adjuvant chemotherapy for active comparator group — 8 cycles of SOX adjuvant chemotherapy will be given to the patients in the active comparator group. The SOX chemotherapy regimen is as follow: S-1 40-60mg Bid, Oral, D1-14, Q21D; Oxaliplatin 130mg/m2, ivgtt, D1, Q21d.
  Arms: Adjuvant Chemotherapy
Drug: Adjuvant chemotherapy for experimental group — 6 cycles of SOX adjuvant chemotherapy will be given to the patients in the experimental group. The SOX chemotherapy regimen is as follow: S-1 40-60mg Bid, Oral, D1-14, Q21D; Oxaliplatin 130mg/m2, ivgtt, D1, Q21d.
  Arms: Adjuvant Chemo-radiotherapy

SUMMARY:
The purpose of this study is to explore the role of adjuvant chemo-radiotherapy in patients with local advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Gastric cancer;
* D2 and R0 resection;
* Pathologically confirmed stage anyT, N+, M0 (AJCC Cancer Staging);
* Karnofsky performance score (KPS) >= 70 or Eastern Cooperative Oncology Group(ECOG) score 0-1;
* Adequate blood counts: White blood cell count ≥3.5 x 109/L Haemoglobin levels ≥100g/L Platelet count ≥100 x 109/L Creatinine levels ≤1.0× upper normal limit（UNL） Urea nitrogen levels ≤1.0× upper normal limit（UNL） Alanine aminotransferase(ALT) ≤1.5× upper normal limit（UNL） Aspartate aminotransferase(AST) ≤1.5× upper normal limit（UNL） Alkaline phosphatase(ALP) ≤1.5× upper normal limit（UNL） Total bilirubin(TBIL) ≤1.5× upper normal limit（UNL）
* No allergic history of 5-Fu or Platinum drugs;
* No history of chemotherapy or other anti-cancer therapy;
* Informed consent should be signed.

Exclusion Criteria:

* GEJ adenocarcinoma
* Concomitant malignancies;(except basocellular carcinoma or in-situ cervical carcinoma)
* Allergic to Fluorouracil or Platinum drugs;
* Concurrent uncontrolled medical condition;
* Known malabsorption syndromes or lack of physical integrity of upper gastrointestinal tract;
* Severe postoperative complications such as anastomotic leakage, etc.;
* Symptoms or history of peripheral neuropathy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Estimated)
Dates: Start 2015-07; Primary Completion 2020-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3 years

SECONDARY OUTCOMES:
Local recurrence free survival | 3 years
Distant metastasis free survival | 3 years
Over all survival | 3 years
Adverse Event | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese academy of medical sciences, Beijing, Beijing Municipality, China